CLINICAL TRIAL: NCT00159926
Title: Does Cleansing of Suction Blood During Cardiac Surgery With Heart and Lung Machine Reduce the Postoperative Inflammatory Response ?
Brief Title: Cleansing of Suction Blood in Cardiac Surgery for Reduced Inflammatory Response
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: For financial and logistical reasons
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Danish Heart Foundation (Other); Copenhagen Hospital Corporation (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 959583153; 961501172; DHF: 03-2-3-35-22109; CHC: 20/fo03
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2008-01-14 (Estimated); Status verified 2007-11

CONDITIONS: Systemic Inflammatory Response Syndrome; Coronary Arteriosclerosis
Keywords: systemic inflammatory response syndrome; coronary artery bypass grafting; cell saver; interleukins; tumor necrosis factor alfa
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome; Coronary Artery Disease | interventions — Operative Blood Salvage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): With cell saver
  Interventions: Procedure: Cell saver
- 2 (Active Comparator): Without cell saver
  Interventions: Procedure: No cell saver

INTERVENTIONS:
Procedure: Cell saver — Cell saver intraoperatively for coronary artery bypass grafting using cardiopulmonary bypass
  Arms: 1
Procedure: No cell saver — Conventional suction for coronary artery bypass grafting using cardiopulmonary bypass
  Arms: 2

SUMMARY:
Cardiac surgery using heart and lung machine produces an inflammatory reaction in the body. This leads in few percent of cases to heart, lung, and kidney disturbances that potentially causes death. White blood cells in contact with the heart and lung machine and external surfaces release mediators partly responsible for this. Blood collected by the suction and the blood remaining in the heart and lung machine after its use, can be cleaned by a cell saver before reinfusion, and this might reduce the inflammatory response.

DETAILED DESCRIPTION:
Introduction

Cardiopulmonary bypass (CPB) during cardiac surgery induces in all patients a systemic inflammatory response syndrome (SIRS) that is more pronounced than for other surgical procedures. Depending on the severity of this, myocardial dysfunction, respiratory failure, renal and neurological dysfunction, coagulation disturbances and impaired liver function might follow. In worst cases this leads to acute respiratory distress syndrome, disseminated intravascular coagulation, multi organ failure, shock and death. The cause is besides the surgical trauma, the passage of the blood through the extra corporal circulation (ECC) and its pumps and oxygenator, hemodilution, hypothermia, heparin and protamine administration, ischemia and reperfusion, and endotoxemia (LPS) as a cause of intestinal ischemia. The ECC is the main cause of immunological activation and leads in severe cases to the so-called post-perfusion syndrome. This is characterised by increased capillary permeability and intercellular fluid, peripheral vasoconstriction, fever, myocardial edema, diffuse cerebral edema and diffuse hemorrhagic diathesis. This syndrome is considered to be a more severe form of SIRS. Even though most patients have no sequelae after CPB, all patients must be considered to be influenced, in varying degree, by SIRS. High levels of pro-inflammatory cytokines (interleukin (IL)-6, IL-8, IL-1a, IL-1b, tumor necrosis factor (TNF) alfa), have generally been associated with adverse events after CPB. Of importance is also LPS from gram-negative intestinal bacteria, translocating to the systemic circulation during ischemia.

Hypothesis

Cleansing of suction blood and the remaining blood in the ECC after termination of CPB, reduces the load of inflammatory cells and mediators in the patients' circulation. This potentially diminishes SIRS with a reduction in postoperative organ dysfunction and morbidity.

Aim

To cleanse suction blood and the remaining blood in the ECC after termination of CPB by means of a cell saver and monitor the influence on inflammatory mediators and the potential clinical benefits.

Outcome measures

Primary: Concentrations of IL-1B, IL-6, IL-8, IL-10, IL-12p70, TNFa, TNF-R1, TNF-R2, PCT and LPS in patient blood: 6, 24 and 72 hours after termination of CPB.

Secondary: Bleeding, need for allogenic blood transfusions and blood products and clinical effect focusing on known complications to cardiac surgery and CPB.

Design

Prospective randomised clinical trial including 40 patients planned for on-pump coronary artery bypass grafting (CABG). n=20 in the trial group (use of cell saver) and n=20 in the control group (no cell saver). No patients receive postoperative autotransfusion of drain blood.

Sample size

Estimation based on comparable studies.

Anaesthesia and surgery

In accordance with current guidelines of the clinic, this includes prophylactic antibiotics (cefuroxime and gentamycin). Cell saver: Medtronic Autolog.

Patient exclusion during the trial

Patients are excluded in cases of autotransfusion of blood not cleansed by the cell saver, for instance in cases of major blood loss.

ELIGIBILITY:
Inclusion Criteria:

* Oral and written informed consent.
* No limits regarding age or ejection fraction.

Exclusion Criteria:

* Off-pump coronary artery bypass grafting
* Redo CABG
* Current infection
* Antibiotic treatment
* S-creatinin > 200 micromol/L
* Antiinflammatory / immuno-modulating treatment: Steroids, immunosuppressive or -stimulating agents (NSAIDs and ASA allowed)
* Liver disease
* Immune disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2003-01; Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
Concentrations of IL-1B, IL-6, IL-8, IL-10, IL-12p70, TNFa, TNF-R1, TNF-R2, PCT and LPS in patient blood. | 6, 24 and 72 hours after termination of CPB.

SECONDARY OUTCOMES:
Bleeding | Intra- and postoperatively
Need for allogenic blood transfusions and blood products | Within submission
Clinical effect focusing on known complications to cardiac surgery and CPB | Within submission

CONTACTS AND LOCATIONS:
Overall Officials: Sune Damgaard, MD, Principal Investigator — Dept. of Cardiothoracic Surgery, Rigshospitalet, Copenhagen; Daniel A Steinbrüchel, Professor, Study Director — Dept. of Cardiothoracic Surgery, Rigshospitalet, Copenhagen
Locations (1):
- Department of Cardiothoracic Surgery, Rigshospitalet, Copenhagen, Denmark